CLINICAL TRIAL: NCT06963268
Title: Validation of the Sentinel Lymph Node Technique in Early-stage Ovarian Cancer (SENTOV II)
Acronym: SENTOV II
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Collaborators: Hospital Universitario La Fe (Other); Hospital Clinic of Barcelona (Other); Hospital Universitario 12 de Octubre (Other); Hospital Universitario La Paz (Other); Hospital General Universitario Gregorio Marañon (Other); Quirón Madrid University Hospital (Other); Hospital of Navarra (Other); Hospital Son Espases (Other); Hospital Universitari de la Vall de Hebron (Unknown); Hospital Universitario Fundación Jiménez Díaz (Other); Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SENTOV II
Record Dates: First submitted 2025-04-30; First posted 2025-05-08 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-04

CONDITIONS: Ovarian Neoplasms
Keywords: Sentinel Node Technique
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: Controlled, prospective, descriptive and not randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Women >18, with confirmed early-stage ovarian cancer, undergoing staging surgery. (Experimental): A 0.2 ml (27 mBq) dose of 99mTc and 0.5 ml (1.25 mg/ml) of ICG is injected subperitoneally in the dorsal or ventral side of the pelvic infundibulum stump, and 0.2 ml (27 mBq) of 99mTc and 1 ml (1.25 mg/ml) of ICG intracervically. Sentinel nodes are located using the auditory signal from the gamma probe and visually via ICG staining with an infrared light system. After 30 minutes, all identified nodes are removed. Deferred histology applies ultra-staging for negative or micrometastatic nodes.
  Interventions: Procedure: Sentinel Node Technique

INTERVENTIONS:
Procedure: Sentinel Node Technique — A 0.2 ml (27 mBq) dose of 99mTc and 0.5 ml (1.25 mg/ml) of ICG is injected subperitoneally in the dorsal or ventral side of the pelvic infundibulum stump, and 0.2 ml (27 mBq) of 99mTc and 1 ml (1.25 mg/ml) of ICG intracervically. Sentinel nodes are located using the auditory signal from the gamma probe and visually via ICG staining with an infrared light system. After 30 minutes, all identified nodes are removed. Deferred histology applies ultra-staging for negative or micrometastatic nodes.

SUMMARY:
This clinical trial investigates the sentinel lymph node (SLN) technique as a less invasive alternative to conventional lymphadenectomy in patients with early-stage ovarian cancer. The primary objective is to evaluate the effectiveness, safety, and diagnostic accuracy of the SLN approach in detecting lymphatic metastases. By assessing its negative predictive value, the study aims to determine whether the SLN technique can reliably replace systematic pelvic and paraaortic lymphadenectomy. If successful, this technique could minimize surgical morbidity, shorten hospitalization stays, and lower complication rates, ultimately improving patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to the performance of any procedure related to the clinical trial.
* Female, 18 years of age or older at the time of inclusion.
* Patients with a histopathological diagnosis of malignant ovarian tumor in a deferred study (any epithelial histology), in apparent early stage FIGO I-II, proposed for staging surgery, or patients with suspected malignant ovarian tumor in apparent early stage FIGO I-II, who will undergo exploratory laparotomy and operative biopsy, and if positive, will undergo staging surgery.

Exclusion Criteria:

* Failure to obtain informed consent or revocation of informed consent.
* Under 18 years of age at the time of inclusion.
* Previous history of vascular surgery on the aorta, vena cava, or pelvic vessels.
* Previous pelvic or paraaortic lymphatic surgery.
* Previous lymphoma.
* Previous abdomino-pelvic tumor.
* Previous allergy to Tc99 or ICG.
* Pregnancy/Breastfeeding.

Patients who have signed informed consent but do not meet all inclusion criteria and none of the exclusion criteria will be considered as selection failures.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Negative predictive value of the sentinel lymph node technique. | Postoperative (30 days +/- 10 days)
  To determine the negative predictive value of the sentinel lymph node technique for detecting lymph node metastases, using pelvic/aortic lymphadenectomy as the Gold Standard.

SECONDARY OUTCOMES:
Concordance of Sentinel Lymph Node Technique vs. Lymphadenectomy | Postoperative (30 days +/- 10 days).
  Evaluate the degree of concordance (sensitivity, specificity, positive predictive value, and diagnostic accuracy) between the sentinel lymph node technique and pelvic/aortic lymphadenectomy (Gold Standard) for detecting lymph node metastasis.
Characterize Sentinel Lymph Node Technique vs. Lymphadenectomy for Metastasis Detection | Intraoperative and postoperative (30 days +/- 10 days).
  Characterize the sentinel lymph node technique for detecting lymph node metastasis using pelvic/aortic lymphadenectomy as the Gold Standard in terms of sensitivity, specificity, positive and negative predictive value, positive and negative likelihood ratios, and effectiveness.
Sample Characterization | Baseline visit and Intraoperative
  Characterize the sample (through collection of baseline characteristics, medical history, tumor markers, intraoperative findings, surgical procedures, and immediate admission data).
Characterize Sentinel Lymph Node Technique Based On Site of Drug Injection | Intraoperative and postoperative (30 days +/- 10 days).
  Characterize the sentinel lymph node technique for detecting lymph node metastasis based on the site of drug injection, using lymphadenectomy as the Gold Standard, in terms of sensitivity, specificity, positive and negative predictive value, positive and negative likelihood ratios, and effectiveness.
Determine Sentinel Lymph Node Procedure Rate | Intraoperative and postoperative (30 days +/- 10 days).
  Determine the sentinel lymph node procedure rate.
Determine the rate of "empty" sentinel lymph node detection. | Postoperative (30 days +/- 10 days).
  Determine the rate of "empty" sentinel lymph node detection.
Determine Pelvic and/or Paraaortic Sentinel Lymph Node Detection Rate | Intraoperative and postoperative (30 days +/- 10 days).
  Determine the detection rate of pelvic and/or paraaortic sentinel lymph nodes.
Identify the anatomical location of the sentinel lymph nodes. | Intraoperative and postoperative (30 days +/- 10 days).
  Identify the anatomical location of the sentinel lymph nodes.
Determine the number of detected lymph nodes. | Intraoperative and postoperative (30 days +/- 10 days).
  Determine the number of detected lymph nodes.
Rate of overstaging with ultrastaging. | Postoperative (30 days +/- 10 days).
  Rate of overstaging with ultrastaging.
Complications related to the sentinel lymph node technique | Intraoperative and postoperative (30 days +/- 10 days).
  Complications related to the sentinel lymph node technique.
Complications related to lymphadenectomy. | Intraoperative and postoperative (30 days +/- 10 days).
  Complications related to lymphadenectomy.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario y Politécnico La Fe, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided